CLINICAL TRIAL: NCT02647073
Title: A Pilot Study to Evaluate the Feasibility of Mobile Monitoring of Vital Signs in Opioid Users
Brief Title: The Mobile Monitoring of Vital Signs in Opioid Users
Acronym: MOVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ongoing issues with the device and software that were provided by the sponsor.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Keith Ahmad, Dr Keith Ahmad, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H15-02986
Record Dates: First submitted 2015-12-22; First posted 2016-01-06 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Opioid Use Disorders
Keywords: Mobile Monitoring; Post-Opioid Consumption; Vital Signs
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile monitoring device arm (Experimental): Canary 01 Mobile Vital Signs Monitoring Device
  Interventions: Device: Canary 01 Mobile Vital Signs Monitoring Device

INTERVENTIONS:
Device: Canary 01 Mobile Vital Signs Monitoring Device — The prototype has several main components, including several commercially available sensors to measure heart rate, respiration, and motion data, an enclosed case containing circuitry for processing and transmitting data, and a mobile phone/system interface to store and transmit data.

SUMMARY:
Opioid dependence and its associated harms are becoming increasingly prevalent in North America, with overdose now being the second leading cause of accidental death in the US. This pilot study will investigate the feasibility of a novel mobile device to monitor vital signs in both opioid-injecting individuals and hospital inpatients who are on high-dose oral opioids. A secondary goal is to explore associations between consumption and changes in vital signs post-injection with the long-term goal of developing a mobile system that will alert clinicians when patients are at risk of overdose so that appropriate interventions can be delivered in time.

DETAILED DESCRIPTION:
1. PURPOSE The purpose of the pilot study is to assess feasibility of a novel device (Canary 01 Mobile Vital Signs Monitoring Device) in individuals who inject opioids and in hospital inpatients who are on high-dose oral opioid medications. The primary objectives are to evaluate if the device can reliably and comfortably be worn for an extended duration of time following opioid consumption and can accurately monitor changes in vital signs (electrocardiogram (ECG), heart rate, respiratory rate) in this clinical population and setting. A secondary purpose of the study is to enrich our understanding of changes in vital signs that occur post-opioid-consumption. The long-term goal of the study is to create a device that will allow clinicians and patients to detect adverse effects of opioid consumption early (i.e. respiratory depression), so that appropriate treatment interventions can be delivered to prevent overdose-related morbidity and mortality.
2. HYPOTHESES The team hypothesizes that the Canary 01 Mobile Vital Signs Monitoring Device will prove to be a feasible and reliable device for monitoring vital signs before and after consumption of opioids, among individuals who inject opioids and among individuals who are on high doses of opioid medication.
3. JUSTIFICATION Opioid medications are key agents for treating acute pain, cancer pain, and are deemed to be essential medicines for pain care by the World Health Organization. However, opioid medications have a serious side effect profile including contributing to delirium, oversedation and respiratory depression in the event of overdose. Between 2005 and 2009, there were 815 deaths related to fentanyl, hydromorphone, morphine and oxycodone in British Columbia. Opioid overdose is now the second leading cause of accidental death in the United States.

   In addition to adverse events, opioids are known to be highly addictive. In Canada, there were an estimated 75,000-125,000 injection drug users (the vast majority of them who injected opioids) as well as approximately 200,000 people with prescription opioid dependence, as of 2012.

   Knowledge gained in this innovative pilot study will inform development of a mobile monitoring device designed to alert clinicians of cardiopulmonary changes indicating opioid overdose in patients, allowing for rapid detection, intervention and administration of potentially life-saving treatment. Ultimately, clinical implementation of this device could lead to a reduction in the substantial morbidity and mortality attributable to opioid-related overdoses.

   In addition, through fulfillment of our secondary objective, this feasibility study will contribute new knowledge regarding changes in cardiopulmonary status associated with use of high opioid doses.
4. OBJECTIVES

Primary Objective To determine whether a mobile monitoring system for specific vital signs (e.g., heart rate and respiratory rate) can be used successfully in the monitoring of opioid dependent individuals.

Specifically, the study team will examine:

1. Participant compliance;
2. Feasibility of specific vital sign data collection, storage, and analysis for participant status assessment; and
3. Clinical utility and overall participant and provider acceptability of mobile monitoring devices

Secondary Objective To document and characterize changes in cardiopulmonary status associated with opioid consumption.

5) RESEARCH METHOD The MOVE study is a single site, three-week feasibility study of individuals who report ongoing/current injection opioid use. Potential study participants will be recruited from the Providence Crosstown Clinic and St. Paul's Hospital. The target enrolment goal is 25.

At the study recruitment sites, potential study candidates will be invited to participate, provide informed consent and complete the Screening Visit (Visit 1) in order to assess eligibility.

Once found to be eligible, individuals recruited at the Crosstown Clinic will complete all other study visits (Visits 2, 3 & 4) at Crosstown Clinic. At Crosstown Clinic, individuals receive managed treatment for opioid dependence with known quantities of drug (e.g. diacetylmorphine, hydromorphone). The clinic is staffed with clinicians who are trained and equipped to deal with any potential opioid overdoses. For hospital inpatients recruited at St. Paul's Hospital, all study visits will occur in hospital.

All participants will be monitored on three separate study visits. At the start of each session and prior to opioid consumption, the study coordinator will assist with placement of two mobile monitoring devices on the study participant to measure specific vital signs:

* Heart rate and ECG monitor: Heart rate and ECG data will be collected with a compact, wireless device with 3 leads that are placed on the participant's chest. The leads are connected to a processor/battery pack unit, approximately the size of a bar of soap.
* Respiratory rate will be collected using Respiratory Inductance Plethysmography (RIP) belts, fastened around the participant's abdomen.
* Activity monitoring: An Inertial Measurement Unit (IMU) (gyro) is incorporated within the device to measure the participant's activity.

At Crosstown Clinic, the participant will receive their managed treatment via self-injection and will be monitored for a total duration of 120 minutes in a clinic room/post-treatment room.

At St. Paul's Hospital, the participant will be administered their dose of oral opioid medications and will be monitored for a duration of 120 minutes ideally at their bedside in their hospital room and always within their hospital ward.

Monitoring devices will be worn for a total duration of 120 minutes. The study coordinator will remain with the participant throughout the observation period. In addition to vital signs data, the study coordinator will complete a activity log documenting all activities that occur during the time that the monitor is in place. In addition any, and all medical treatments and/or interventions administered during this time will be recorded by members of the study team.

Data from the mobile monitors will be transmitted via Bluetooth to a smart phone, and then securely transmitted to the study database. Transmitted data will be coded with the participant's study identification code only and will not contain any protected health information and will not be utilized for any clinical decision-making.

It is important to highlight that data collected from the mobile monitoring device will solely be used for research and will not serve any clinical decision-making purpose.

All participants will be discharged from the study at Visit 4. Participants will be offered addiction treatment referrals if requested.

Safety data will be collected up to 30 days following the last study visit and follow-up of any serious adverse events will continue until resolution.

THE MOBILE VITAL SIGNS MONITORING DEVICE

The prototype has several main components, including several commercially available sensors to measure heart rate, respiration, and motion data, an enclosed case containing circuitry for processing and transmitting data, and a mobile phone/system interface to store and transmit data.

Data is collected from respiratory bands, ECG electrodes, and an accelerometer. The safety of individual sensor components has been evaluated previously by respective manufacturers and all are currently available for commercial purposes. Two respiratory bands, worn on the thorax and abdomen, will measure patterns and changes in participant breathing patterns. Although not yet implemented, outputs such as breaths per minute could be extracted from the data file by using peak finding or frequency analysis software in future. Four ECG electrodes placed on the participant's thorax and abdomen will record analog voltage changes that correspond to the electrical potential difference that occur during the cardiac cycle (i.e. heartbeat). The electrodes are configured in a 3-lead setup, with three signal electrodes and a driven electrode. In the unlikely event that the device malfunctions, Analog Devices ECG chips with a current-limiting protection circuit have been used to optimize participant safety, as per manufacturer specifications. The 3-axis analog accelerometer is sampled at 10 Hz, and used to denote activity and motion artefacts that may influence ECG and respiratory data.

These sensors are attached to a custom printed circuit board (PCB) and a Bluetooth module inside a 3D printed case. The PCB holds two microprocessors needed for the system: the PIC16LF1618 and the Broadcom Wireless Internet Connectivity for Embedded Devices (WICED) Smart. The WICED Smart communicates sensor data to the mobile phone using Bluetooth Low Energy (BLE). The case holds the circuit boards and a 3.7 V lithium-ion battery; the circuit boards are screwed into a separate compartment inaccessible to patients.

The circuit board processes and sends the data to a phone application. Data is then transferred wirelessly to a Standardized Query Language (SQL) database. Within this database, each data point is associated with a timestamp and patient Identification (ID), allowing for multiple patients' data to be stored in the same SQL database. Finally, the battery included in the case has been tested to last for two days of continuous use.

6) STATISTICAL ANALYSIS

Descriptive statistics, including the mean, standard deviation, median and 95% confidence intervals of the mean for continuous variables, and frequency distribution for categorical variables will be produced for participant demographics and baseline characteristics.

STATISTICAL METHODS FOR PRIMARY AND SECONDARY OUTCOMES

As this is a feasibility study, more complex statistical analyses are not planned.

EXPLORATORY ANALYSES

Biometric data collected before and after opioid consumption will be compiled and used to construct preliminary simulation models of average changes in heart rate and respiratory rate following consumption of high dose opioids. Ultimately, the goal of these modeling exercises will be to develop a clinical algorithm to be used with the mobile signs monitoring device to determine thresholds of risk and levels of therapeutic intervention required at each threshold.

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 64 years of age, inclusive;
2. Current and ongoing injection drug use with opioids OR hospitalized inpatients under the care of the St. Paul's Hospital Addiction Medicine Consult Team with current and ongoing use of high dose oral opioid medications;
3. Current and past history of an opioid use disorder;
4. Ability to communicate in English; and
5. Ability to provide written informed consent and comply with study procedures.

Exclusion Criteria:

1. Inability to understand study procedures due to changed health and/or mental status;
2. Chest circumference greater than 115 cm;
3. Women who are pregnant or breastfeeding
4. Has a pacemaker or automatic cardioverter defibrillator (AICD) in situ;
5. Diagnosed with atrial fibrillation;
6. Have other medical devices (i.e. insulin pump) that precludes the use of the device;
7. Allergies or skin conditions that preclude the use of adhesive electrodes; and
8. Any other condition that, in the judgment of the investigator, presents a contraindication to study participation.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Estimated); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Participant compliance: Proportion of participants who wear the device | For Visit 2, Visit 3 and Visit 4 (>100 minutes per 120minute session). Visits will take place over an average of 3 weeks
  Proportion of participants who wear the device for >100 minutes per 120 minute session as reported by participants and observed by the study coordinator/nurse.
Feasibility: Proportion of participant sessions with continuous transmission of vital signs data | For Visit 2, Visit 3 and Visit 4( >100 minutes per 120 minute session). Visits will take place over an average of 3 weeks
  Proportion of participant sessions with continuous transmission of vital signs data for >100 minutes per 120 minute session
Clinical utility | through study completion
  Compiled scores and summary data (means, medians, ranges) from participant & clinician usability surveys.

SECONDARY OUTCOMES:
Study retention and drop-out rates | Through study completion, an average of 3 weeks per participant
Premature device removal event counts and rates (participant or clinician initiated); | Through study completion, an average of 3 weeks per participant.
Reliability of device as measured by artefact and transmission failure rates; | Through study completion, an average of 3 weeks per participant
Characterization of physiological changes following opioid consumption; | For Visit 2, Visit 3 and Visit 4 for 120 minutes. Visits will take place over an average of 3 weeks
For a subset of participants enrolled in the hospital, accuracy of data recorded by the device in comparison to data collected by bedside monitoring equipment | For Visit 2, Visit 3 and Visit 4 at various time points per 120 minute session.Visits will take place over an average of 3 weeks per participant.
  HR and RR

CONTACTS AND LOCATIONS:
Overall Officials: Keith Ahamad, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Crosstown Community Clinic, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No